CLINICAL TRIAL: NCT03671889
Title: Assessment of Safety and Efficacy of ExAblate Blood-Brain Barrier Disruption for the Treatment of Patients With Probable Alzheimer's Disease
Brief Title: ExAblate Blood-Brain Barrier (BBB) Disruption for the Treatment of Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: AL002
Record Dates: First submitted 2018-08-03; First posted 2018-09-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Alzheimer Syndrome; Magnetic Resonance guided Focal Ultrasound (MRgFUS); Blood-Brain Barrier; ExAblate
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Subjects who meet study eligibility will undergo treatment procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Blood Brain Barrier (BBB) Disruption (Experimental): ExAblate Model 4000 Type 2.0 System
  Interventions: Device: Blood Brain Barrier (BBB) Disruption

INTERVENTIONS:
Device: Blood Brain Barrier (BBB) Disruption — Focal Ultrasound (FUS) involves the application of acoustic energy at low frequencies from over 1000 individual transducers into distinct targets to induce BBB disruption.
  Other Names: ExAblate Neuro

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the ExAblate Model 4000 Type 2.0 System as a tool to disrupt the blood-brain barrier (BBB) in patients with probable Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to evaluate the safety and efficacy of BBB disruption using the ExAblate Model 4000 Type 2.0 (220 kHz) system. Patients with diagnosis of Probable Alzheimer's Disease may qualify for a clinical trial to have three serial ExAblate BBB disruption procedures in specific areas in the brain. This study will be conducted at up to 8 sites in the United States and will enroll up to 30 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female between 50-85 years of age
2. Probable Alzheimer's Disease (AD)
3. If taking concurrent Alzheimer's medication, has been on the medication for at least 2 months with a stable dose for at least 3 months
4. Able to communicate sensations during the ExAblate MRgFUS procedure
5. Ambulatory

Exclusion Criteria:

1. MRI Findings
2. Presence of unknown or MR unsafe devices anywhere in the body
3. Significant cardiac disease or unstable hemodynamic status
4. Relative contraindications to ultrasound contrast agent or PET amyloid tracer
5. History of a bleeding disorder
6. History of liver disease
7. Known cerebral or systemic vasculopathy
8. Significant depression and at potential risk of suicide
9. Any contraindications to MRI scanning
10. Any contraindication to lumbar puncture for collection of cerebral spinal fluid
11. Untreated, uncontrolled sleep apnea
12. History of seizure disorder or epilepsy
13. Severely Impaired renal function
14. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device or in any other type of medical research
15. Chronic pulmonary disorders
16. Positive human immunodeficiency virus (HIV)
17. Known apolipoprotein E allele (ApoE4) homozygosity

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Device and procedure related adverse events | 5 years
  Rate of adverse events following each treatment through end of study

OTHER OUTCOMES:
BBB Disruption and Closure | Immediately after the end of each ExAblate treatment and 24 hours post treatment
  MR images post-procedure to verify that the BBB was disrupted and subsequently closed within 24 hours.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Delray Medical Center & Florida Atlantic University, Delray Beach, Florida
  - Broward Health Medical Center & The University of Florida, Fort Lauderdale, Florida
  - University of Florida Health Shands, Gainesville, Florida
  - Baptist Health South Florida & Florida International University, Miami, Florida
  - Advent Health, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Weill Cornell Medicine, New York, New York
  - The Ohio State University -Wexner Medical Center, Columbus, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - West Virginia University Rockefeller Neuroscience Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta RI, Carpenter JS, Mehta RI, Haut MW, Wang P, Ranjan M, Najib U, D'Haese PF, Rezai AR. Ultrasound-mediated blood-brain barrier opening uncovers an intracerebral perivenous fluid network in persons with Alzheimer's disease. Fluids Barriers CNS. 2023 Jun 16;20(1):46. doi: 10.1186/s12987-023-00447-y. PMID 37328855
- [Derived] Rezai AR, Ranjan M, Haut MW, Carpenter J, D'Haese PF, Mehta RI, Najib U, Wang P, Claassen DO, Chazen JL, Krishna V, Deib G, Zibly Z, Hodder SL, Wilhelmsen KC, Finomore V, Konrad PE, Kaplitt M; Alzheimer's Disease Neuroimaging Initiative. Focused ultrasound-mediated blood-brain barrier opening in Alzheimer's disease: long-term safety, imaging, and cognitive outcomes. J Neurosurg. 2022 Nov 4;139(1):275-283. doi: 10.3171/2022.9.JNS221565. Print 2023 Jul 1. PMID 36334289
- [Derived] Mathew AS, Gorick CM, Price RJ. Multiple regression analysis of a comprehensive transcriptomic data assembly elucidates mechanically- and biochemically-driven responses to focused ultrasound blood-brain barrier disruption. Theranostics. 2021 Oct 11;11(20):9847-9858. doi: 10.7150/thno.65064. eCollection 2021. PMID 34815790
- [Derived] Mehta RI, Carpenter JS, Mehta RI, Haut MW, Ranjan M, Najib U, Lockman P, Wang P, D'haese PF, Rezai AR. Blood-Brain Barrier Opening with MRI-guided Focused Ultrasound Elicits Meningeal Venous Permeability in Humans with Early Alzheimer Disease. Radiology. 2021 Mar;298(3):654-662. doi: 10.1148/radiol.2021200643. Epub 2021 Jan 5. PMID 33399511